CLINICAL TRIAL: NCT06624059
Title: A Phase I-III, Multicenter Study Evaluating the Efficacy and Safety of Multiple Therapies in Cohorts of Patients With Resectable Stage I-III Non-Small Cell Lung Cancer, Selected According to Biomarker Status
Brief Title: A Study to See How Well and How Safely Different Treatments Work in a Group of Participants With Non-Small Cell Lung Cancer (NSCLC)
Acronym: HORIZON 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO43249
Record Dates: First submitted 2024-10-01; First posted 2024-10-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort B1 (Experimental): Participants will receive alectinib in combination with platinum-based chemotherapy for up to 4 cycles (cycle length = 3 weeks), followed by alectinib monotherapy for up to 5 years.
  Interventions: Drug: Alectinib; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Cohort B2 (Experimental): Participants will receive alectinib and platinum-based chemotherapy for up to 3 cycles (cycle length = 3 weeks) prior to surgery, and alectinib monotherapy after surgery for up to 5 years after surgery.
  Interventions: Drug: Alectinib; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Alectinib — Cohort B1: participants will receive oral alectinib twice daily (BID) for up to 5 years.
  Cohort B2: Participants will receive oral alectinib BID for 3 cycles (cycle length = 3 weeks) prior to surgery, and for up to 5 years after surgery.
Drug: Cisplatin — Cohort B1: Participants will receive intravenous (IV) cisplatin on Day 1 of each cycle for up to 4 cycles (cycle length = 3 weeks).
  Cohort B2: Participants will receive IV cisplatin on Day 1 of each cycle for up to 3 cycles (cycles length = 3 weeks) prior to surgery.
Drug: Carboplatin — Cohort B1: Participants will receive IV carboplatin on Day 1 of each cycle for up to 4 cycles (cycle length = 3 weeks).
  Cohort B2: Participants will receive IV carboplatin on Day 1 of each cycle for up to 3 cycles (cycle length = 3 weeks) prior to surgery.
Drug: Pemetrexed — Cohort B1: Participants will receive IV pemetrexed on Day 1 of each cycle for up to 4 cycles (cycle length = 3 weeks).
  Cohort B2: Participants will receive IV pemetrexed on Day 1 of each cycle for up to 3 cycles (cycle length = 3 weeks) prior to surgery.

SUMMARY:
The objective of this study is to evaluate the efficacy and/or safety of multiple therapies in patients with early-stage resectable NSCLC. Cohort B1 is a phase II cohort that will evaluate the safety, and efficacy of alectinib in combination with up to four cycles of platinum-based chemotherapy in the adjuvant setting post complete surgical resection. Cohort B2 is a phase II cohort that will evaluate the efficacy and safety of perioperative alectinib in combination with chemotherapy in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria Cohort B1:

* Complete resection of the primary NSCLC with negative margins
* Confirmed stage II to select stage IIIB (T3N2) NSCLC of non-squamous (adenocarcinoma) histology
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1

Inclusion Criteria Cohort B2:

* Evaluation by the operating attending surgeon and involved medical oncologist prior to study enrollment to verify study eligibility for complete surgical resection with curative intent
* Pathologically and/or histologically confirmed Stage II-IIIA and IIIB (T3N2 only) NSCLC of non-squamous (adenocarcinoma) histology

Inclusion Criteria Cohorts B1 and B2:

* Documented ALK fusion

Exclusion Criteria Cohort B1:

* NSCLC of squamous or mixed histology regardless of the presence of an ALK mutation
* Prior exposure to any systemic anti-cancer therapy

Exclusion Criteria Cohort B2:

* NSCLC of squamous or mixed histology regardless of the presence of an ALK mutation
* Known sensitivity to any component of alectinib, pemetrexed, cisplatin, or carboplatin
* Prior exposure to any systemic anti-cancer therapy

Exclusion Criteria Cohorts B1 and B2:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-06-13 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Cohort B1: Incidence, type, and severity of adverse events (AEs) with onset up to 28 days after the last dose of chemotherapy | Up to 28 days after the last dose of chemotherapy treatment (up to 4 cycles, cycle length = 3 weeks)
Cohort B2: Investigator-assessed pathologic complete response (inv-pCR) | At the time of surgical resection (approximately weeks 14-17)

SECONDARY OUTCOMES:
Cohort B1: Investigator-assessed disease-free survival (DFS) | From initiation of study treatment to the first documented recurrence of disease or new primary NSCLC or death from any cause, whichever occurs first (up to approximately 5 years)
Cohort B1: Overall survival (OS) | From initiation of study treatment to death from any cause (up to approximately 8 years)
Cohort B1: Incidence, type, and severity of AEs with onset up to 28 days after the last dose of study treatment | From first dose to up to approximately 5 years
Cohort B1: Time to first onset of selected AEs | From first dose to up to approximately 5 years
Cohort B1: Change from baseline in target safety parameters | From first dose to up to approximately 5 years
Cohort B2: Investigator-assessed major pathological response (inv-MPR) | At the time of surgical resection (approximately weeks 14-17)
Cohort B2: Pathologic complete response (pCR) by independent review | At the time of surgical resection (approximately weeks 14-17)
Cohort B2: Major pathologic response (MPR) by independent review | At the time of surgical resection (approximately weeks 14-17)
Cohort B2: Investigator-assessed overall response rate (ORR) | Up to approximately Week 17
Cohort B2: Investigator-assessed event-free survival (EFS) | From first treatment to the first documented disease progression that prevents surgery, local or distant disease recurrence, or death from any cause (up to approximately 5 years)
Cohort B2: Overall Survival (OS) | From initiation of study treatment to death from any cause (up to approximately 8 years)
Cohort B2: Incidence, severity, and type of AEs | From first dose up to approximately 5 years
Cohort B2: Change from baseline in target safety parameters | From first dose to up to approximately 5 years
Cohort B2: Frequency of surgery completion, defined as participants who have successfully completed surgery without treatment-related delays (> 60 days) from the last dose of neoadjuvant treatment | At the time of surgical resection (approximately weeks 14-17)
Cohort B2: Length of treatment-related surgical delays, incidence of operative and post-operative complications, and/or reasons for surgical cancellations | Approximately weeks 14-24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo, Brazil
- RedSalud Vitacura, Santiago, Chile
- China (5):
  - Beijing Cancer Hospital, Beijing
  - The third people's hospital of Chengdu, Chengdu
  - Guangdong General Hospital, Guangzhou
  - Jinhua municipal central hospital, Jinhua
  - Yunnan Cancer Hospital, Kunming
- Institut Gustave Roussy, Villejuif, France
- Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia, Perugia, Umbria, Italy
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing